CLINICAL TRIAL: NCT04106700
Title: Venous Thromboembolism Prophylaxis With Apixaban in Transplant Eligible Patients With Newly Diagnosed Multiple Myeloma Receiving Induction Therapy With an Immunomodulatory-based Regimen
Brief Title: Prophylaxis With Apixaban in Transplant Eligible Patients With Multiple Myeloma Receiving Induction Therapy With IMiDs
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low recruitment
Sponsor: Instituto de Investigacion Sanitaria La Fe (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APIXABAN
Record Dates: First submitted 2019-09-20; First posted 2019-09-27 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2020-06

CONDITIONS: Venous Thromboembolism
Keywords: Multiple Myeloma; Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism; Multiple Myeloma | interventions — apixaban

STUDY DESIGN:
Intervention Model Description: Clinical trial with a single arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Apixaban (single arm) (Experimental)
  Interventions: Drug: Apixaban 2.5 MG

INTERVENTIONS:
Drug: Apixaban 2.5 MG — Apixaban will be started simultaneously with anti myeloma treatment on day 1 of cycle 1 of VTD, and continues for 4 to 6 months depending on the number of induction cycles administered to the patient

SUMMARY:
Interventional, no-randomized, open-label, and single arm multicentre study of apixaban for the prevention of thromboembolic events during induction therapy in transplant-eligible patients with newly diagnosed multiple myeloma who receive bortezomib, thalidomide, and dexamethasone (VTD) during the induction phase of therapy prior to autologous stem cell transplantation (ASCT). The current study is designed to evaluate the efficacy and safety of apixaban during the induction period. Efficacy will be defined as a composite endpoint of acute symptomatic proximal and distal deep venous thrombosis, pulmonary embolism, VTE related deaths, and acute ischemic stroke.

DETAILED DESCRIPTION:
This study is designed to test the efficacy and safety of the oral anti factor Xa apixaban 2.5 mg given twice daily as a prophylaxis of VTE in transplant-eligible patients with multiple myeloma during the induction therapy with VTD.

Induction therapy prior to ASCT will consist in no less than 4 and no more than 6 cycles of VTD, depending on treatment response. Duration of each cycle is 4 weeks if there is not any disease or treatment-related complication; therefore, treatment duration will be around 4-6 months. Daily Prophylaxis with apixaban will continue up to a maximum of 14 days after the last dose of thalidomide. In addition, there will be an additional observation period of 14 (± 7) days, starting the day after the last dose of study medication (until 28 days after the end of the last cycle of VTD).

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Subjects must have documented newly diagnosed symptomatic multiple myeloma requiring front-line treatment.
* Patients should be considered transplant-eligible
* Subjects will receive front-line induction therapy with a triplet regimen consisting of bortezomib, thalidomide and dexamethasone (VTD).
* To enter to the study at the same time of start anti myeloma induction therapy.
* Ages eligible for study: 18 to 70 years.
* Subjects must have an Eastern Cooperative Oncology Group (ECOG) performance status score ≤2.

Exclusion Criteria:

* Patients with the diagnosis of plasma cell leukemia, Waldenström macroglobulinemia, POEMS syndrome or amyloidosis of light chain.
* Patients with smouldering multiple myeloma or monoclonal gammopathy of undeterminated significance.
* Patients considered non-transplant-eligible.
* Grade ≥2 of peripheral neuropathy.
* Prior history of documented any venous thromboembolism and arterial thrombosis event
* Active or high risk of bleeding.
* Need for on-going anticoagulant or antiplatelet treatment.
* Contraindication of anticoagulant prophylaxis
* Uncontrolled hypertension: systolic blood pressure >200 mmHg and/or diastolic blood pressure >100 mmHg.
* HIV, HBV or HCV-positive active.
* Expected survival <6 months.
* Weight <40 Kg.
* Low platelet count (<50 x109/L).
* ALT >3x UNL, bilirubin >2x ULN.
* Creatinine clearance <30 mL/min.
* Women of childbearing potential who are unwilling to use an acceptable method of contraception.
* Women of childbearing potential who are pregnant or breastfeeding.
* Women with a positive pregnancy test on enrollment, prior to investigational product administration.
* Administration of any investigational drug currently or within 30 days prior to planned enrollment into this study.
* Subjects unwilling or unable to comply with study medication instructions or study procedures (e.g. bilateral lower extremity venous ultrasonography).
* Known allergies to ingredients contained in apixaban.
* Use of any contraindicated medications with apixaban (see section 5.4.1).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-04-12 (Actual); Primary Completion 2020-08-26 (Actual); Study Completion 2020-10-05 (Actual)

PRIMARY OUTCOMES:
Venous thromboembolism (VTE)- related death | Cycle 1 Day 1 (each cycle is 28 days. Treatment will finish on cycle 4 or 6. Treatment with Apixaban will continue until 14 days after cycle 4/6)
  i.e. death for which VTE can not be excluded as a cause
Venous thromboembolism (VTE)- related death | Cycle 2 Day 1 (each cycle is 28 days. Treatment will finish on cycle 4 or 6. Treatment with Apixaban will continue until 14 days after cycle 4/6)
  i.e. death for which VTE can not be excluded as a cause
Venous thromboembolism (VTE)- related death | Cycle 3 Day 1 (each cycle is 28 days. Treatment will finish on cycle 4 or 6. Treatment with Apixaban will continue until 14 days after cycle 4/6)
  i.e. death for which VTE can not be excluded as a cause
Venous thromboembolism (VTE)- related death | Cycle 4 Day 1 (each cycle is 28 days. Treatment will finish on cycle 4 or 6. Treatment with Apixaban will continue until 14 days after cycle 4/6)
  i.e. death for which VTE can not be excluded as a cause
Venous thromboembolism (VTE)- related death | Cycle 5 Day 1(each cycle is 28 days. Treatment will finish on cycle 4 or 6. Treatment with Apixaban will continue until 14 days after cycle 4/6)
  i.e. death for which VTE can not be excluded as a cause
Venous thromboembolism (VTE)- related death | Cycle 6 Day 1 (each cycle is 28 days. Treatment will finish on cycle 4 or 6. Treatment with Apixaban will continue until 14 days after cycle 4/6)
  i.e. death for which VTE can not be excluded as a cause
Venous thromboembolism (VTE)- related death | Cycle 4 Day 29 (each cycle is 28 days. Treatment will finish on cycle 4 or 6. Treatment with Apixaban will continue until 14 days after cycle 4/6)
  i.e. death for which VTE can not be excluded as a cause
Venous thromboembolism (VTE)- related death | Cycle 6 Day 29 (each cycle is 28 days. Treatment will finish on cycle 4 or 6. Treatment with Apixaban will continue until 14 days after cycle 4/6)
  i.e. death for which VTE can not be excluded as a cause
Venous thromboembolism (VTE)- related death | Cycle 4 Day 43 (each cycle is 28 days. Treatment will finish on cycle 4 or 6. Treatment with Apixaban will continue until 14 days after cycle 4/6)
  i.e. death for which VTE can not be excluded as a cause
Venous thromboembolism (VTE)- related death | Cycle 6 Day 43 (each cycle is 28 days. Treatment will finish on cycle 4 or 6. Treatment with Apixaban will continue until 14 days after cycle 4/6)
  i.e. death for which VTE can not be excluded as a cause
Venous thromboembolism (VTE)- related death | 14 days after last dose of apixaban
  i.e. death for which VTE can not be excluded as a cause
Symptomatic deep-vein thrombosis (DVT) | Cycle 1 Day 1 (each cycle is 28 days. Treatment will finish on cycle 4 or 6. Treatment with Apixaban will continue until 14 days after cycle 4/6)
  Lower extremity DVT: erythema (redness of the skin), warmth, pain, swelling, tenderness
Symptomatic deep-vein thrombosis (DVT) | Cycle 2 Day 1 (each cycle is 28 days. Treatment will finish on cycle 4 or 6. Treatment with Apixaban will continue until 14 days after cycle 4/6)
  Lower extremity DVT: erythema (redness of the skin), warmth, pain, swelling, tenderness
Symptomatic deep-vein thrombosis (DVT) | Cycle 3 Day 1 (each cycle is 28 days. Treatment will finish on cycle 4 or 6. Treatment with Apixaban will continue until 14 days after cycle 4/6)
  Lower extremity DVT: erythema (redness of the skin), warmth, pain, swelling, tenderness
Symptomatic deep-vein thrombosis (DVT) | Cycle 4 Day 1 (each cycle is 28 days. Treatment will finish on cycle 4 or 6. Treatment with Apixaban will continue until 14 days after cycle 4/6)
  Lower extremity DVT: erythema (redness of the skin), warmth, pain, swelling, tenderness
Symptomatic deep-vein thrombosis (DVT) | Cycle 5 Day 1 (each cycle is 28 days. Treatment will finish on cycle 4 or 6. Treatment with Apixaban will continue until 14 days after cycle 4/6)
  Lower extremity DVT: erythema (redness of the skin), warmth, pain, swelling, tenderness
Symptomatic deep-vein thrombosis (DVT) | Cycle 6 Day 1 (each cycle is 28 days. Treatment will finish on cycle 4 or 6. Treatment with Apixaban will continue until 14 days after cycle 4/6)
  Lower extremity DVT: erythema (redness of the skin), warmth, pain, swelling, tenderness
Symptomatic deep-vein thrombosis (DVT) | Cycle 4 Day 29 (each cycle is 28 days. Treatment will finish on cycle 4 or 6. Treatment with Apixaban will continue until 14 days after cycle 4/6)
  Lower extremity DVT: erythema (redness of the skin), warmth, pain, swelling, tenderness
Symptomatic deep-vein thrombosis (DVT) | Cycle 6 Day 29 (each cycle is 28 days. Treatment will finish on cycle 4 or 6. Treatment with Apixaban will continue until 14 days after cycle 4/6)
  Lower extremity DVT: erythema (redness of the skin), warmth, pain, swelling, tenderness
Symptomatic deep-vein thrombosis (DVT) | Cycle 4 Day 43 (each cycle is 28 days. Treatment will finish on cycle 4 or 6. Treatment with Apixaban will continue until 14 days after cycle 4/6)
  Lower extremity DVT: erythema (redness of the skin), warmth, pain, swelling, tenderness
Symptomatic deep-vein thrombosis (DVT) | Cycle 6 Day 43 (each cycle is 28 days. Treatment will finish on cycle 4 or 6. Treatment with Apixaban will continue until 14 days after cycle 4/6)
  Lower extremity DVT: erythema (redness of the skin), warmth, pain, swelling, tenderness
Symptomatic deep-vein thrombosis (DVT) | 14 days after last dose of apixaban
  Lower extremity DVT: erythema (redness of the skin), warmth, pain, swelling, tenderness
Pulmonary embolism (PE) | Cycle 1 Day 1 (each cycle is 28 days. Treatment will finish on cycle 4 or 6. Treatment with Apixaban will continue until 14 days after cycle 4/6)
  Pleuritic chest pain, dyspnea (shortness of breath), cough, hemoptysis (expectoration of blood or blood-stained sputum), syncope (fainting), lightheadedness/dizziness, tachypnea (rapid breathing), tachycardia (fast heart rate).
Pulmonary embolism (PE) | Cycle 2 Day 1 (each cycle is 28 days. Treatment will finish on cycle 4 or 6. Treatment with Apixaban will continue until 14 days after cycle 4/6)
  Pleuritic chest pain, dyspnea (shortness of breath), cough, hemoptysis (expectoration of blood or blood-stained sputum), syncope (fainting), lightheadedness/dizziness, tachypnea (rapid breathing), tachycardia (fast heart rate).
Pulmonary embolism (PE) | Cycle 3 Day 1 (each cycle is 28 days. Treatment will finish on cycle 4 or 6. Treatment with Apixaban will continue until 14 days after cycle 4/6)
  Pleuritic chest pain, dyspnea (shortness of breath), cough, hemoptysis (expectoration of blood or blood-stained sputum), syncope (fainting), lightheadedness/dizziness, tachypnea (rapid breathing), tachycardia (fast heart rate).
Pulmonary embolism (PE) | Cycle 4 Day 1 (each cycle is 28 days. Treatment will finish on cycle 4 or 6. Treatment with Apixaban will continue until 14 days after cycle 4/6)
  Pleuritic chest pain, dyspnea (shortness of breath), cough, hemoptysis (expectoration of blood or blood-stained sputum), syncope (fainting), lightheadedness/dizziness, tachypnea (rapid breathing), tachycardia (fast heart rate).
Pulmonary embolism (PE) | Cycle 5 Day 1 (each cycle is 28 days. Treatment will finish on cycle 4 or 6. Treatment with Apixaban will continue until 14 days after cycle 4/6)
  Pleuritic chest pain, dyspnea (shortness of breath), cough, hemoptysis (expectoration of blood or blood-stained sputum), syncope (fainting), lightheadedness/dizziness, tachypnea (rapid breathing), tachycardia (fast heart rate).
Pulmonary embolism (PE) | Cycle 6 Day 1 (each cycle is 28 days. Treatment will finish on cycle 4 or 6. Treatment with Apixaban will continue until 14 days after cycle 4/6)
  Pleuritic chest pain, dyspnea (shortness of breath), cough, hemoptysis (expectoration of blood or blood-stained sputum), syncope (fainting), lightheadedness/dizziness, tachypnea (rapid breathing), tachycardia (fast heart rate).
Pulmonary embolism (PE) | Cycle 4 Day 29 (each cycle is 28 days. Treatment will finish on cycle 4 or 6. Treatment with Apixaban will continue until 14 days after cycle 4/6)
  Pleuritic chest pain, dyspnea (shortness of breath), cough, hemoptysis (expectoration of blood or blood-stained sputum), syncope (fainting), lightheadedness/dizziness, tachypnea (rapid breathing), tachycardia (fast heart rate).
Pulmonary embolism (PE) | Cycle 6 Day 29 (each cycle is 28 days. Treatment will finish on cycle 4 or 6. Treatment with Apixaban will continue until 14 days after cycle 4/6)
  Pleuritic chest pain, dyspnea (shortness of breath), cough, hemoptysis (expectoration of blood or blood-stained sputum), syncope (fainting), lightheadedness/dizziness, tachypnea (rapid breathing), tachycardia (fast heart rate).
Pulmonary embolism (PE) | Cycle 4 Day 43 (each cycle is 28 days. Treatment will finish on cycle 4 or 6. Treatment with Apixaban will continue until 14 days after cycle 4/6)
  Pleuritic chest pain, dyspnea (shortness of breath), cough, hemoptysis (expectoration of blood or blood-stained sputum), syncope (fainting), lightheadedness/dizziness, tachypnea (rapid breathing), tachycardia (fast heart rate).
Pulmonary embolism (PE) | Cycle 6 Day 43 (each cycle is 28 days. Treatment will finish on cycle 4 or 6. Treatment with Apixaban will continue until 14 days after cycle 4/6)
  Pleuritic chest pain, dyspnea (shortness of breath), cough, hemoptysis (expectoration of blood or blood-stained sputum), syncope (fainting), lightheadedness/dizziness, tachypnea (rapid breathing), tachycardia (fast heart rate).
Pulmonary embolism (PE) | 14 days after last dose of apixaban
  Pleuritic chest pain, dyspnea (shortness of breath), cough, hemoptysis (expectoration of blood or blood-stained sputum), syncope (fainting), lightheadedness/dizziness, tachypnea (rapid breathing), tachycardia (fast heart rate).
Asymptomatic proximal DVT as detected by systematic compression ultrasound | Cycle 4 Day 43 (each cycle is 28 days. Treatment will finish on cycle 4 or 6. Treatment with Apixaban will continue until 14 days after cycle 4/6)
  Diagnostic assessment of DVT. Presence of any one of the following will be considered diagnostic for the presence of DVT:
  1. New or previously undocumented non-compressibility of one or more proximal venous segments (popliteal vein or higher) of the legs on compression ultrasound.
  2. Constant intraluminal filing defect(s) in two or more views on contrast venography in one or more venous segments in the legs or pelvis, or involving the inferior vena cava.
Asymptomatic proximal DVT as detected by systematic compression ultrasound | Cycle 6 Day 43 (each cycle is 28 days. Treatment will finish on cycle 4 or 6. Treatment with Apixaban will continue until 14 days after cycle 4/6)
  Diagnostic assessment of DVT. Presence of any one of the following will be considered diagnostic for the presence of DVT:
  1. New or previously undocumented non-compressibility of one or more proximal venous segments (popliteal vein or higher) of the legs on compression ultrasound.
  2. Constant intraluminal filing defect(s) in two or more views on contrast venography in one or more venous segments in the legs or pelvis, or involving the inferior vena cava.

SECONDARY OUTCOMES:
Major bleeding event | Cycle 1 Day 1, Cycle 2 Day 1, Cycle 3 Day 1, Cycle 4 Day 1, Cycle 5 Day 1, Cycle 6 Day 1, Cycle 4/ 6 Day 29, Cycle 4/6 Day 43, Day 14 after end of treatment (each cycle is 28 days. Treatment with Apixaban will continue until 14 days after cycle 4 or 6)
  Defined as a bleeding event that is acute clinically overt bleeding accompanied by one or more of the following:
  * A decrease in hemoglobin (Hb) of 2 g/dL or more over a 24-hour period.
  * A transfusion of 2 or more units of packed red blood cells.
  * Bleeding that occurs in at least one of the following critical sites: intracranial, intra-spinal, intraocular (within the corpus of the eye; thus, a conjunctival bleed is not an intraocular bleed), pericardial, an operated joint and requires re-operation or intervention, intramuscular with compartment syndrome, retroperitoneal.
  * Bleeding that is fatal.
Clinically relevant non-major bleeding event | Cycle 1 Day 1, Cycle 2 Day 1, Cycle 3 Day 1, Cycle 4 Day 1, Cycle 5 Day 1, Cycle 6 Day 1, Cycle 4/ 6 Day 29, Cycle 4/6 Day 43, Day 14 after end of treatment (each cycle is 28 days. Treatment with Apixaban will continue until 14 days after cycle 4 or 6)
  Defined as a bleeding event that is:
  * Acute clinically overt bleeding.
  * Does not satisfy additional criteria required for the bleeding event to be defined as a major bleeding event and meets at least one of the following criteria:
  * Epistaxis: need to medical attention from a physician or visits an emergency room, requires an intervention, persists for 5 minutes or more.
  * Gastrointestinal bleed: vomit containing frank blood or coffee ground material which tests positive for blood, endoscopically confirmed bleeding, frank blood per rectum or melena stools.
  * Hematuria: overt spontaneous bleeding, bleeding persists for 24 hours or more after instrumentation.
  * Bruising/ecchymosis: any bruise, which is assessed as "unusual".
  * Hematoma: presence of a hematoma is demonstrated radiographically, and a drop-in hemoglobin is present with no external evidence of bleeding.
  * Hemoptysis: expectoration of blood or blood-stained sputum.
Fatal Bleeding Event | Cycle 1 Day 1, Cycle 2 Day 1, Cycle 3 Day 1, Cycle 4 Day 1, Cycle 5 Day 1, Cycle 6 Day 1, Cycle 4/ 6 Day 29, Cycle 4/6 Day 43, Day 14 after end of treatment (each cycle is 28 days. Treatment with Apixaban will continue until 14 days after cycle 4 or 6)
  Defined as a bleeding event that determines is the primary cause of death or contributes directly to death.
Liver injury event | Cycle 1 Day 1, Cycle 2 Day 1, Cycle 3 Day 1, Cycle 4 Day 1, Cycle 5 Day 1, Cycle 6 Day 1, Cycle 4/ 6 Day 29, Cycle 4/6 Day 43, Day 14 after end of treatment (each cycle is 28 days. Treatment with Apixaban will continue until 14 days after cycle 4 or 6)
  Potential or suspected cases of liver injury including but not limited to liver test abnormalities (elevation of ALT, AST, GGT, alkaline phosphatase and total bilirrubin), jaundice, hepatitis or cholestasis events.
Serious adverse events | Cycle 1 Day 1, Cycle 2 Day 1, Cycle 3 Day 1, Cycle 4 Day 1, Cycle 5 Day 1, Cycle 6 Day 1, Cycle 4/ 6 Day 29, Cycle 4/6 Day 43, Day 14 after end of treatment (each cycle is 28 days. Treatment with Apixaban will continue until 14 days after cycle 4 or 6)
  A Serious Adverse Event is any untoward medical occurrence that:
  * Results in death.
  * Is life-threatening (defined as an event in which the subject was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe).
  * Requires inpatient hospitalization or prolongation of existing hospitalization
  * Results in persistent or significant disability/incapacity.
  * Is a congenital anomaly/birth defect.
  * Is an important medical event (defined as a medical event(s) that may require medical intervention to prevent one of a serious outcome listed above).
  * Overdose.
  * Second primary malignancies.
Symptomatic DVT or PE occurring during the 90 days of follow-up period | Day +90 follow-up
  Symptomatic DTV or PE as defined aforementioned, assessed 90 days after the last dose of the study drug.
Death occurring during the 90 days of follow-up period | Day +90 follow-up
  All cause of mortality occurring during the 90 days after the last dose of the study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Javier de la Rubia, Study Director — Hospital Doctor Peset; Samuel Romero, Principal Investigator — Hospital Universitario y Politecnico La Fe
Locations (4):
- Spain (4):
  - Hospital Clinico Universitario, Valencia
  - Hospital Universitario Doctor Peset, Valencia
  - Hospital Universitario y Politécnico La Fe, Valencia
  - Hospital General Universitario, Valencia

IPD SHARING:
Plan to Share IPD: No